CLINICAL TRIAL: NCT05374746
Title: Evaluation of Parents' Knowledge and Attitudes About Signs and Symptoms of Infant Teething
Brief Title: Evaluation of Parents' Knowledge About Infant Teething
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Assoc. prof. dr, Istanbul University
Other Study IDs: 2021/34
Record Dates: First submitted 2022-05-08; First posted 2022-05-16 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Signs and Symptoms
Keywords: Signs and Symptoms; Tooth Eruption; Child
MeSH Terms: conditions — Signs and Symptoms; Exanthema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Many children may have general disorders such as sleep disorders, lack of appetite, fever, diarrhea, vomiting, coughing and respiratory problems during tooth eruption.These symptoms usually occur in6-36 monthchildren. The emergent symptoms don't affect not only children but also parents try to find solutions to these symptoms. Parents' knowledge level and their way trying finda solution to these symptoms may differ.

The aim of this study is to evaluate the perceptions of parents towards the teething signs and symptoms of their children aged 6-36 months-old.As a result of the research, it is aimed to organize educational programs for families by increasing the knowledge level of parents about teething symptoms.

DETAILED DESCRIPTION:
The study is being carried out in Istanbul University Department of Pediatric Dentistry, period between September 2021 - August 2022 following the ethics committee approval 2021/34. Patient parents are informed about the study and the written informed consents are obtained from parents of all participants included in the study. The questionnaireis conducted face-to-face. Parents with children between 6-36 months-oldwho has been applying to the Department of Pedodontics at Istanbul University Faculty of Dentistry are asked to complete the questionnaire consisting of 55 questions.

Questionnaire:

8 questions to find out the sociodemographic characteristics, 6 questions to find out the characteristics of the baby 6 questions to find out the general knowledge about children's teething 23 questions to find outthe teething symptoms that are seen in their babies 3 questions to find out the timing of the symptoms 9 questions to find out the parents practices in managing teething problems. Questionnaire responses are being recorded. The answers will be evaluated with statistical analyses. Detailed analyses of responses will be carried out according to sociodemographic characteristics, family structures and educational levels of parents.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Parents who have 6-36 months old child
* Presence of parents who can adequately answer the questionnaire questions

Exclusion Criteria:

* Not willing to participte in the study
* Parents with no children for the specific age group
* In case of not being able to answer the questionnaire questions from the parents

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents with 6 month to 3 year children
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
A questionnaire form covering questions regarding evaluation of parents' perception towards the teething signs and symptoms | 1 Year
  The tool which is used a questionnaire form covering questions regarding sociodemographic characteristics, characteristics of the baby, general knowledge about children's teething, teething symptoms that are seen in their babies, timing of the symptoms, parents practices in managing teething problems.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Tuna, Prof.Dr, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No